CLINICAL TRIAL: NCT04753892
Title: An Immune Challenge Model Using gp41 3Sm Peptide in Healthy Human Adults to Characterise B Cell Responses to a Model Virus-neutralizing Antibody-inducing Motif in Health Versus Chronic Viral Infection
Brief Title: 3Sm Challenge Model Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Minka Therapeutics (Unknown); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21HH6540
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): The 3Sm peptide is conjugated to a mutant diphtheria carrier protein (CRM197) and the resulting challenge agent (3SM2-G-CRM197) will be mixed with a squalene adjuvant before intramuscular administration at Months 0, 1, 2 and 4, at a dosage of 32 micrograms of 3SM2-G-CRM197 and 9.7 micrograms of adjuvant.
  Interventions: Other: 3SM2-G-CRM197 with squalene adjuvant

INTERVENTIONS:
Other: 3SM2-G-CRM197 with squalene adjuvant — Immune challenge agent

SUMMARY:
The 3Sm challenge study is a small clinical study in eight healthy volunteers who will be injected with a protein which includes a short portion ('3Sm peptide') which is derived from a part (the '3S region') of the coat protein of HIV. The researchers believe that the 3Sm peptide might trigger an immune response which includes rare antibodies able to neutralise a wide range of different strains of HIV. The results will be useful in guiding the development of future vaccines against HIV, and other diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged between 18 and 55 years on the day of screening.
2. Willing and able to provide written informed consent.
3. Available for all follow-up visits for the duration of the study.
4. Entered into and obtained clearance from The Over volunteering Prevention System (TOPS) database (to avoid impact of any co-administered investigational products or treatments on our outcomes).
5. If female and of childbearing potential, willing to use a highly effective method of contraception from screening until a minimum of 6 weeks after the last immunogen challenge. Periodic abstinence (calendar, symptothermal and post-ovulation methods) and withdrawal are not acceptable methods of contraception.
6. If male and not sterilised, willing to avoid impregnating female partners through the use of condoms or sexual abstinence from screening until a minimum of 6 weeks after the last immunogen challenge, unless female partners are using a highly effective method during the same time period.
7. Registered with a GP in the UK prior to enrolment into the study.
8. Willing to grant authorised persons access to his/her trial-related medical record and GP records either directly or indirectly
9. Willing to avoid all vaccines from within 4 weeks before the first immunogen challenge through to 4 weeks after the final challenge, with the exception of seasonal influenza vaccine which may be given more than 7 days before or after the experimental immunogen, and deployed COVID-19 vaccine which may be given 14 days before or after the experimental immunogen (and at least 28 days is encouraged). It is recommended that participants have an up to date vaccination status for any required immunisations.

Exclusion Criteria:

1. Pregnant or lactating
2. History of any physical, medical, psychological or other condition, clinically significant laboratory, vital sign or examination finding at screening, or use of any medications which, in the opinion of the investigators, would interfere with the study objectives or participant's safety. This includes where there is a history of active disease requiring a clinically significant recent or planned investigation or change in treatment, including cardiac, respiratory, endocrine, metabolic, autoimmune, liver, neurological, oncological, psychiatric, immunosuppresive/immunodeficient or other disorders. Individuals with mild/moderate, well-controlled co-morbidities, of those that are no longer deemed clinically active or clinically significant by the investigator are allowed.
3. History of anaphylaxis or angioedema.
4. History of severe or multiple allergies to drugs or pharmaceutical agents.
5. History of severe local or general reaction to vaccination defined as:

   1. local: extensive, indurated redness and swelling involving most of the arm, not resolving within 72 hours
   2. general: fever ≥39.5 °C within 48 hours; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
6. Previous receipt of an investigational vaccine or immunogen based on HIV envelope.
7. Detection of antibodies to HIV.
8. Detection of antibodies to Hepatitis C.
9. Unable to read and/or speak English to a fluency level adequate for the full comprehension of study procedures and consent.
10. Participation in another study, or treatment with an investigational drug within 28 days of screening, which in the opinion of the investigator would interfere with study objectives or compromise the participant's safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Serum titres of 3Sm antibodies | From Month 0 to Month 6
  ELISA read-outs
Frequency of 3Sm secreting B cells in peripheral blood | From Month 0 to Month 6
  ELISpot read-outs

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Pollock, MD, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial Clinical Research Facility, London, Please Select..., United Kingdom

IPD SHARING:
Plan to Share IPD: No